CLINICAL TRIAL: NCT07014111
Title: Fight Fatigue: A Progressive Muscle Relaxation and Walking Intervention to Reduce Fatigue in Adults With ESKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mary Hannan, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY2025-0281; R34AT012770 (NIH)
Record Dates: First submitted 2025-05-23; First posted 2025-06-10 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-06

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fight Fatigue (Experimental): Combined progressive muscle relaxation and walking (increasing step count) 12-week intervention that consists of education/training followed by text messages
  Interventions: Behavioral: Fight Fatigue
- Attention Control (Active Comparator): End-stage kidney disease education, followed by text messages (over 12 weeks)
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: Fight Fatigue — Combined progressive muscle relaxation and walking (increasing step count) 12-week intervention that consists of education/training followed by text messages.
  Arms: Fight Fatigue
Other: Attention Control — End-stage kidney disease education
  Arms: Attention Control

SUMMARY:
Fight Fatigue is evaluating the feasibility and acceptability of a combined progressive muscle relaxation and walking intervention to reduce fatigue for adults with end-stage kidney disease receiving in-center hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ESKD diagnosis and receiving hemodialysis for at least 3 months
* Can read and speak English
* Fatigue measured via visual analogue scale, score ≥4 over the last week
* Able to stand and walk one block
* Has a cell phone that can receive text messages

Exclusion Criteria:

* Patient's nephrologist refuses for them to participate
* Unstable angina
* Unstable pulmonary disease or pulmonary symptoms that preclude participation
* Lower-extremity amputation without prosthetic (BKA, AKA) -Orthopedic or neurologic condition that would preclude walking or tensing/releasing of muscles-
* Cognitive impairment that, in the judgement of the research team, precludes trial participation
* Participation in the formative phase of the development of Fight Fatigue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Baseline to week 12
  Recruitment metrics (enrolled/invited)
Feasibility of retention | Baseline to week 12
  Retention in the study from baseline to week 12
Acceptability | End of study (Week 12)
  Participant rating of acceptability (e.g., enjoyable, easy to understand) via Likert scale questions and open ended questions
Adherence to the study protocol | Baseline to week 12
  Adherence to the intervention measured with adherence to step counts, number/duration of accesses on the study-specific website, and adherence to study procedures as evaluated with number of text messages read/sent messages read.

OTHER OUTCOMES:
Fatigue | Baseline to week 12
  FACIT-Fatigue measure

CONTACTS AND LOCATIONS:
Locations (1):
- UI Health/University of Illinois Chicago, Chicago, Illinois, United States